CLINICAL TRIAL: NCT00715377
Title: Anticholinergic Burden in Schizophrenia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient subject accrual
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Ariel Graff, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 118/2007
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder; Delusional Disorder; Psychotic Disorders
Keywords: benztropine; Anticholinergic antiparkinsonian agents; antipsychotics; elderly population; side-effects
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Schizophrenia, Paranoid | interventions — Benztropine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Benztropine

INTERVENTIONS:
Drug: Benztropine — Patients aged ≥ 50 years suffering from a primary psychotic disorder treated with a SGA and benztropine concomittantly at any dose steadily for at least 3 months will be eligible to participate in this study. The dose of benztropine will be reduced by 0.5mg per week. During this 8-week study period, extrapyramidal symptoms will be assessed on a weekly basis. The clinical assessments will be repeated 8 weeks after the initial assessments.

SUMMARY:
Anticholinergic antiparkinsonian agents often cause side-effects including cognitive impairment, dry mouth, and constipation while they diminish antipsychotic-induced parkinsonian symptoms. The introduction of second generation antipsychotics (SGA) brought fewer neurological side effects. However, anticholinergic coprescription rates are still as high as 12-65% in patients on SGA that are much higher than the incidence of EPS reported in clinical trials (3-20%). This apparently discrepancy is likely explained, in part, by the established tradition of routine use of this medications. Older patients are particularly sensitive to anticholinergic side-effects due to age-related changes in pharmacokinetics and pharmacodynamics. In this study, we will examine the safety and benefits of reducing the dose of a frequently prescribed anticholinergics, benztropine, on cognitive function, extrapyramidal symptoms, and psychotic symptoms in older subjects with a primary psychotic disorder.

DETAILED DESCRIPTION:
Anticholinergic antiparkinsonian agents (AAAs) are frequently prescribed in patients with a primary psychotic disorder either to treat or prevent the emergence of antipsychotic induced extrapyramidal symptoms (EPS). Second generation antipsychotics (SGAs) are by definition associated with fewer neurological side effects. This would be expected to be associated with a lower use of AAAs. However, in a recent prescription survey, Park and colleagues found that while the rate of concomitant use of antiparkinsonian agents dropped by 9.2% in patients with schizophrenia after changing their antipsychotic from typical antipsychotics to SGAs, 30% of prescriptions for SGAs included a concomitant antiparkinsonian agent. This is consistent with the results of other cross-sectional surveys demonstrating anticholinergic co-prescription rates of 12 - 65% in patients treated with SGA. These high rates are remarkable especially when one considers that the incidence of EPS reported in past clinical trials using SGAs (3 - 20%) is much lower than this reported co-prescription rate. This apparent discrepancy is likely explained, in part, by the established tradition of prophylactic (or routine) use of AAAs for patients starting antipsychotic drugs.

The adverse effects of AAAs are well known, and are particularly significant clinically in the elderly, who are at high risk of cognitive impairment with AAAs. Anticholigergic effects have been reported to impair cognitive function both globally as well as in specific domains, including memory and executive functioning. The association between anticholinergic activity and cognitive performance are also strongly supported by recent studies measuring serum anticholinergic activity (SAA).

Furthermore, in addition to their well-known side effects such as dry mouth, blurred vision, and constipation, they have also been reported to increase the risk of tardive kinesia and have been claimed to have a negative impact on the clinical efficacy of antipsychotic drugs.

In view of these adverse effects, the World Health Organization has discouraged the prophylactic use of AAAs, and a careful risk-benefit analysis is necessary for each individual patient. Since most cases of antipsychotic-induced EPS present within 11 weeks of initiation of antipsychotic treatment or a dosage increase, a trial of AAA taper and discontinuation has been recommended following 3 months of regular AAA treatment. These recommendations emerged prior to the widespread use of SGAs, and one might expect that successful discontinuation of concomitant AAAs would be higher for SGAs than conventional antipsychotics. AAA discontinuation trials for conventional antipsychotics have been inconsistent, with some studies reporting favorable outcomes and others reporting re-emergence of EPS. More recently Mori et al reported a favorable outcome following AAA discontinuation for both cognition and EPS in patients maintained on chlorpromazine, risperidone, or haloperidol in mixed age population with schizophrenia.

The only study of AAA discontinuation in older patients with schizophrenia also reported improved cognitive function in a sample of 21 elderly inpatients with schizophrenia. However, this study did not include extrapyramidal symptoms, psychopathology, or other side effects from AAAs as outcome measures. Furthermore, improvement in cognitive function reported in this study could be attributed to practice effects: the Alzheimer's Disease Assessment Scale-Cognitive subscale was administered at intervals of 10 days - though the learning effects of this scale have not been studied in patients with schizophrenia.

Older patients with schizophrenia would be expected to be particularly sensitive to side effects to both antipsychotics and AAAs due to age-related changes in pharmacokinetics and pharmacodynamics. However, in view of the well known adverse effects of AAAs in the elderly, use of anticholinergic drugs is specifically included in the 2002 criteria for potentially inappropriate medication used in older adults. This may be especially relevant to older patients with schizophrenia since their cognitive function is already impaired as a function of the dual effects of age-related decline and the cognitive difficulties inherent to the psychotic illness itself. Concomitant use of AAAs would be expected to lead to a further decline in their cognitive and social functioning.

We therefore propose an open-label prospective trial to assess the feasibility of reducing the dose of a frequently prescribed AAA at our Centre, benztropine, in older subjects with a primary psychotic disorder on SGAs using validated assessment scales and methods. In order to quantify the anticholinergic burden in these patients before and after AAA dose reduction, serum anticholinergic activity will be also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age of 50 and older
* DSM-IV/SCID diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or psychotic disorder NOS
* Having been treated with benztopine at a steady daily dose of 3 mg or less for at least three months
* Having been treated with risperidone, quetiapine, olanzapine, or clozapine at a steady dose for at least two weeks.
* Willingness to provide consent for investigator to communicate with their physician of record regarding their participation in the study.

Exclusion Criteria:

* Unstable physical illness or clinically significant neurological disorder
* A history of severe or life-threatening dystonia
* Presence of EPS defined as a total score of 7 or more or a score of 3 or more on any individual item on the SAS at baseline
* Positive urine drug screen for illegal drugs

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
percentage of participants who successfully withdraw from anticholinergic antiparkinsonian agents. | at the end of the study

SECONDARY OUTCOMES:
effect of reducing the dose of benztropine on EPS and anticholinergic side-effects including cognitive impairments. | intermittent

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Graff, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health — http://www.camh.net/research